CLINICAL TRIAL: NCT02443129
Title: Swept Source Enhanced Depth Imaging Optical Coherence Tomography (SS-EDI-OCT) and Study of the Retina, Choroid and Sclera in Health and Disease
Brief Title: Swept Source Enhanced Depth Imaging Optical Coherence Tomography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 185/14
Record Dates: First submitted 2015-03-01; First posted 2015-05-13 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Retina, Choroid, Sclera

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- control group (Experimental): 18-99 year old male + female
  Intervention:
  DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- mydramide only (Experimental): Patients in the clinics undergoing pupil dilation
  Intervention:
  Tropicamide instillation to both eyes DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- mydramide and ephrine 10% (Experimental): Patients in the clinics undergoing pupil dilation
  Intervention:
  Tropicamide and ephrine 10% instillation to both eyes DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- All patients presenting with RD (Experimental): Patients with retinal detachment
  Intervention:
  RD surgery DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- Impact of previous grid treatment (Experimental): Patients after grid laser
  Intervention:
  DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- Effect of glaucoma medications (Experimental): Patients requiring new intraocular presssur (IOP)-lowering treatment Patients with long-term IOP-lowering treatment
  Intervention:
  If needed, start of new IOP-lowering treatment DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- Effect of arteritic/non-arteritic AION (Experimental): About 180 living patients diagnosed at ShaareZedek with anterior ischemic optic neuropathy (AION).
  Longitudinal arm with newly diagnosed patients for 2 years follow-up
  Intervention:
  DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- NVAMD poorly responsive to Rx (Experimental): Patients with neovascular age-related macular degeneration and epiretinal membreane/vitreomacular traction who do not respond to first course of Avastin
  Intervention:
  DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon
- Retrospective analysis (Experimental): All patients pictured with DRI-OCT
  Intervention:
  DRI-1 Swept source OCT, Atlantis, Topcon
  Interventions: Device: DRI-1 Swept source OCT, Atlantis, Topcon

INTERVENTIONS:
Device: DRI-1 Swept source OCT, Atlantis, Topcon — Fundus imaging

SUMMARY:
The investigators would be interested in applying the enhanced depth imaging technique to swept source optical coherence tomography, by modifying the acquisition protocol. Doing so, the investigators hope to improve the visualization of the choroid and perhaps even of the sclera.

DETAILED DESCRIPTION:
A structurally and functionally normal choroidal vasculature is essential for retinal function. The status of the choroid appears to be a crucial determinant in the pathogenesis of diseases such as age-related choroidal atrophy, myopic chorioretinal atrophy, central serous chorioretinopathy, chorioretinal inflammatory diseases, and tumors.

The in vivo structure of the choroid in health and disease is incompletely visualized with traditional imaging modalities, including indocyanine green angiography and ultrasonography.

Optical coherence tomography (OCT) is an established medical imaging technique that uses light to capture micrometer-resolution, three-dimensional images from within optical scattering media. OCT is based on low-coherence interferometry. Nowadays, it is essential for managing retinal conditions.

Unfortunately, standard spectral domain optic coherence tomography (SD-OCT) is of limited use in imaging choroidal morphology.

A modification to the standard technique, termed enhanced depth imaging optical coherence tomography (EDI-OCT), is able to image the choroid with better clarity using commercial SD-OCTs.

With the advent of enhanced depth imaging optical coherence tomography (EDI-OCT), detailed visualisation of the choroid in vivo has been made possible possible. Measurements of choroidal thickness (CT) have also enabled new directions in research to study normal and pathological processes within the choroid.

However, EDI-OCT has its own limitations: the outer choroidal border cannot always be visualized and choroidal details sometime lack clarity.

A new generation of OCTs has been made available, based on swept-source technology.

Swept source OCT (SS-OCT) has been shown to be more precise than spectral domain EDI-OCT in measuring choroidal thickness.

Our department is now using two OCTs, one is a SD- OCT (Canon HS-100), the other one a SS- OCT (Topcon DRI Atlantis).

The investigators would be interested in applying the EDI technique to SS- OCT, by modifying the acquisition protocol. Doing so, the investigators hope to improve the visualization of the choroid and perhaps even of the sclera.

This modification is based on the technique described by Spaide for SD-OCT.

From the patient's perspective, it only involves spending more time fixing the green stimulus (about 4 minutes instead of 2, in order to follow the swept-source EDI protocol in addition to standard swept source).

ELIGIBILITY:
Inclusion Criteria:

* Ability to sit for OCT

Exclusion Criteria:

* Media opacities precluding fundus view

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Difference in chorio-retinal depth and morphology between healthy and diseased subjects | 2 years